CLINICAL TRIAL: NCT05277389
Title: Addressing Socioeconomic Disparities in Post-stroke Upper-extremity Disability Through the Development of an Accessible, New Tool
Brief Title: New Tool to Enhance Post-stroke Upper Extremity Disability
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Claire Honeycutt, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00002440
Record Dates: First submitted 2022-02-14; First posted 2022-03-14 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator): Individuals in this group will practice object manipulation tasks without the START (Startle Adjuvant Rehabilitation Therapy) intervention
  Interventions: Other: Sham Control
- START (Experimental): Individuals in this group with practice object manipulation tasks with the START condition (startling acoustic stimuli applied during 33% of trials)
  Interventions: Other: START - Startle Adjuvant Rehabilitation Therapy

INTERVENTIONS:
Other: START - Startle Adjuvant Rehabilitation Therapy — Application of startling acoustic stimuli during practice of movement task
  Arms: START
Other: Sham Control — Practice of Movement task without START
  Arms: Control

SUMMARY:
Individuals with low socioeconomic status (SES) are more likely to have a stroke, more disabled at 3 months, and less likely to be independently ambulatory. Individuals with low SES struggle to adhere to physician guidelines because of 1) increased disability leaves patients ineligible or unable to tolerate therapy, and 2) poor access to quality care i.e., lack of transportation to therapy. To reduce post-stroke disparity in low SES groups, society must invest in development of novel tools that make therapy more accessible. For the past 5 years, the PI has been developing Startle Adjuvant Rehabilitation Therapy (START), a tele-enabled, low-cost treatment to improve upper-extremity therapy outcomes in individuals with stroke - in particular individuals with severe-to-moderate stroke. START is the application of a startling, acoustic stimulus (via headphones) which increases the intensity of practice, particularly in severe patient populations. START is adjuvant, meaning it does not replace clinical practice but instead enhances current evidence-based treatments. Objective: the investigators seek to determine if START can be used to enhance functionally relevant movement of the upper extremity. Preliminary data: Individuals with severe-to-moderate disability from a stroke completed a remotely delivered, 3-day training of object manipulation with START. Box and Blocks, which was targeted during training, demonstrated a large increase under START (+47.1%) compared to Control (+3.3%). Modified functional reach was also increased under START (+8.9%) compared to Control (+1.1%). Impairment also decreased under START (Upper-Extremity-Fugl-Meyer: +8.6%) resulting in subject-reported increase in arm function both in quantity (Motor Activity Log: +26.2%) and quality (+20.2%). These results indicate that START can be deployed remotely and may prove a valuable, adjuvant tool to enhance functional upper extremity movement. The investigators propose to perform a Phase 1 clinical trial on a larger cohort of 58 subjects, with a longer, 5-day training with the goal of establishing that START can 1) enhance functional movement of the upper extremity and 2) generate sustainable changes that impact quality of life. Impact: This proposal is significant because it tests a tool that has the potential to directly target the causes leading to disparity of care for individuals with low SES. A third (34%) of 6.5 million people in the U.S. with stroke are on Medicaid or uninsured. Our best evidence-based therapies (e.g., high-intensity, CIMT) and our emerging rehabilitation technologies (e.g., TMS, robotics) are inaccessible to our minority and low SES populations. START addresses disparity because it 1) targets individuals with severe disability, which disproportionally affects low SES and minority groups, and 2) is tele-enabled eliminating transportation which 60% of individuals with low SES report as a barrier to care. If successful, this study will set the stage for larger trials to establish 1) the effectiveness of START to be incorporated into traditional therapy and as well as patient compliance, adherence, and tolerance - particularly in low SES groups.

DETAILED DESCRIPTION:
Individuals with low socioeconomic status (SES) are more likely to have a stroke and more likely to have severe upper extremity dysfunction following that stroke. Patients from low SES backgrounds receive less out-patient care, are discharged more quickly, and are less likely to receive evidence-based, guideline recommended care. The mechanisms underlying disparity in treatment are multifaceted but a crucial contributor is individuals with low SES struggle to adhere to clinician guidelines because of 1) poor access to quality care - 60% of individuals with low SES report lack of transportation as a barrier to care, 2) increased severity requires high-intensity/ high-dose therapy which is not fully covered by traditional copay models or Medicaid/Medicare which have caps on therapy costs. To reduce post-stroke disparity in low SES groups, society needs to invest in the development of novel tools that make therapy more accessible or society runs the risk of furthering the inequities that leave our poor and minority populations unable to participate in daily life and return to work.

The PI has been developing Startle Adjuvant Rehabilitation Therapy (START), a tele-enabled, low-cost treatment to improve therapy outcomes in individuals with stroke - in particular individuals with severe stroke. START is the application of a startling, acoustic stimulus (via headphones) administered in conjunction with traditional therapy. Distinct from other auditory treatments (e.g. metronome), START represents endogenous activation of the cortico-reticular system that increases the intensity of practice leading to faster therapy outcomes, particularly in severe stroke. START increases the intensity of muscle activity i.e., more frequent activity onset, larger amplitude (2-3-fold higher than maximum voluntary capacity), and faster onsets. START is adjuvant, meaning it does not replace clinical practice but instead enhances current evidence-based treatments. As START can be administered safely with a cellphone and headphones (often already available to patients), patients can continue to practice at home safely without therapist supervision.

OBJECTIVE: Determine if START can be used to enhance functionally relevant movement of the upper extremity. In our preliminary data, individuals with severe-to-moderate disability from a stroke completed a remotely delivered, 3-day training with START. Box and Blocks had a large increase under START (+47.1%) compared to Control (+3.3%). The Modified Functional Reach Test also increased under START (+8.9%) compared to Control (+1.1%). Impairment decreased under START (Upper-Extremity-Fugl-Meyer: +8.6%) resulting in subject-reported increase in arm function both in quantity (Motor Activity Log: +26.2%) and quality (+20.2%).

These results indicate that START can be deployed remotely and may prove a valuable, adjuvant tool to enhance functional upper extremity movement. The investigators propose to perform a Phase 1 clinical trial on a larger cohort of 58 subjects, with a longer, 5-day training, and more rigorous assessment of function with the goal of establishing that START can 1) enhance functional movement of the upper extremity and 2) generate sustainable changes that impact quality of life.

The investigation team is uniquely positioned to pursue these objective. The team made up experts in START, upper-extremity post-stroke disability, engineering including app development (Claire Honeycutt, PhD, PI), physical therapy, high-intensity training, focus in severe stroke (Pamela Bosch, DPT, PhD, Co-I), occupational therapy, remote delivery/telehealth, rater fidelity, randomized controlled trials (Veronica Rowe, PhD, OTR/L, Co-I). Finally, a data analytics/statistics consultant (Venn Ravichandran, PhD). Together, the investigators will explore the following aims.

Aim 1: To establish that START can increase functional paretic limb usage, the investigators will perform a randomized controlled trial assessing the impact of START on therapy outcomes. The investigators will perform a stratified, parallel-group, double-blind, randomized controlled trial with individuals with severe-moderate stroke (UEFM 0-42/66; MAS 0-4/4) - with recruitment focused on individuals with low SES. Following baseline assessment, subjects will receive training consisting of 5 consecutive days of training focusing on object manipulation. Subjects will either receive therapy with START or without (Control). Outcome measures will be: % change in paretic arm impairment (Upper-Extremity Fugl-Meyer: FMA-UE), spasticity (modified Ashworth: MA & modified Tradieu Scales: MTS), function (Action Research Arm Test: ARAT), patient reported Quality of life (stroke impact scale: SIS), functional independence (modified Rankin Scale: mRS), and arm function (Motor Activity Log: MAL). H1: Training with START will increase paretic arm function (ARAT) and self-reported arm function (MAL) compared to training without START.

Aim 2: To establish that START generates sustainable functional changes that impact quality of life, the investigators will re-assess upper-extremity function and self-reported quality of life at one-month. All outcome measures (FMA-UE, MA, MTS, ARAT, SIS, mRS, MAL) will be re-administered one-month post training. H2: START gains will be retained more than Control and retention will be associated with higher quality of life measures (e.g., SIS, MAL) one-month post-START training.

IMPACT: This proposal is significant because it tests a tool that has the potential to directly target the causes leading to disparity of care for individuals with low SES. A third (34%) of 6.5 million people in the U.S. with stroke are on Medicaid or uninsured. Our best evidence-based therapies (e.g., high-intensity, CIMT) and our emerging rehabilitation technologies (e.g., TMS, robotics) are inaccessible to our minority and low SES populations. START addresses disparity because it 1) targets individuals with severe disability, which disproportionally affects low SES and minority groups, and 2) is tele-enabled eliminating transportation. If successful, this study will set the stage for larger trials to establish 1) the effectiveness of START to be incorporated into traditional therapy and as well as patient compliance, adherence, and tolerance - particularly in low SES groups.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old
2. Capacity to provide informed consent
3. Cerebral stroke at least 6 months prior to testing
4. Presence of upper extremity impairment associated with stroke
5. Corrected pure tone threshold (octave frequencies 250- 4000 Hz) norms for their age and gender27,28 NOTE: Audiometry data will be collected for all participants by lab personnel trained by an audiologist in a sound-attenuated booth. We expect that ~30% of participants will use hearing aids; we will not exclude these individuals but rather include hearing aid use as a covariate in analyses.

Exclusion Criteria:

1. Severe concurrent medical problems (e.g. uncontrolled cardiorespiratory impairment)
2. Acute/painful condition/injury of upper extremity/spine that interfere with ability to participate.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Tempe, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 12/20/22 - 12/15/23 Locations: Medical clinics, community fliers, gyms, events related to stroke, online community groups and members.
Pre-assignment Details: 3 participants withdrawn for reasons as follow: 1 safety concern pertaining to mobility, 1 upper extremity pain, 1 illness before 1st session
Period: Overall Study
Arm/Group | Control | START
Started | 11 | 10
Completed | 10 | 6
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | START | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (13) | 48 (19) | 54 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 10 | 6 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 1 | 2
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Action Research Arm Test (ARAT) Total Score From Baseline to Post-Intervention
Description: The Action Research Arm Test (ARAT) assesses upper extremity function, specifically arm and hand motor abilities, in individuals with neurological conditions. The test evaluates grasp, grip, pinch, and gross movement through 19 standardized tasks. Each task is scored from 0 (no movement) to 3 (normal movement), yielding four subscale scores (Grasp, Grip, Pinch, Gross Movement) that are summed to compute a total score. The total score ranges from 0 to 57, with higher scores indicating better upper extremity function. Subscale ranges are: Grasp (0-18), Grip (0-12), Pinch (0-18), and Gross Movement (0-9). The outcome measure reports the change in the total ARAT score from baseline to post-intervention, with positive values reflecting improved function. Scores are reported as units on a scale.
Time Frame: Time from Baseline to Post-intervention (1 week intervention, 1 month post intervention - total 5 weeks time frame)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control | START
Number analyzed (Participants) | 11 | 10
Units on a scale | 0.72 (1.737292) | 0 (2.692582)

2. Primary Outcome: Retention in Action Research Arm Test (ARAT)
Description: as for outcome 1
Time Frame: Comparing baseline to one-month post (1 month post intervention - total 5 weeks time frame)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control | START
Number analyzed (Participants) | 11 | 10
Units on a scale | 1 (1.603567) | -0.666667 (3.204164)

3. Primary Outcome: Change in Motor Activity Log (MAL) Amount of Use Score From Baseline to Post-Intervention
Description: The Motor Activity Log (MAL) assesses arm use in daily activities post-stroke. The Amount of Use subscale (0-5) rates 30 tasks; higher scores mean more use. Total score averages task scores (0-5). Change in total score is reported. Units on a scale. MAL was taken at baseline and then at one-month post intervention.
Time Frame: Time from Baseline to Post-intervention (1 week intervention, 1 month post intervention - total 5 weeks time frame)
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Control | START
Number analyzed (Participants) | 11 | 10
units on scale | -2.045455 (12.02384) | 0.388889 (5.085382)

4. Primary Outcome: Retention in Motor Activity Log (MAL)
Description: The Motor Activity Log (MAL) assesses arm use in daily activities post-stroke. The Amount of Use (AOU) subscale (0-5) rates 30 tasks; higher scores indicate more use. The total score sums the 30 AOU task scores, ranging from 0 to 150. Units on a scale.
Time Frame: Retention of measure comparing baseline to one-month
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Control | START
Number analyzed (Participants) | 11 | 10
units on scale | 5.0625 (8.174164) | 12.75 (21.731889)

5. Secondary Outcome: Change in Upper Extremity Fugl Meyer (UEFM) Baseline to Post-intervention
Description: The Fugl-Meyer Assessment for Upper Extremity (FMA-UE) evaluates motor function post-stroke via 33 tasks. Total score (0-66) sums subscales: shoulder/arm (0-36), wrist/hand (0-24), coordination (0-6). Higher scores indicate better function. Units on a scale. FMA-UE was taken at baseline and then at one-month post intervention.
Time Frame: Time from Baseline to Post-intervention (1 week intervention, 1 month post intervention - total 5 weeks time frame)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | START
Number analyzed (Participants) | 11 | 10
units on a scale | 0.090909 (3.935849) | 1.555556 (3.574602)

6. Secondary Outcome: Retention of Upper Extremity Fugl Meyer From End Training to One-month Post
Description: The Fugl-Meyer Assessment for Upper Extremity (FMA-UE) evaluates motor function post-stroke via 33 tasks. Total score (0-66) sums subscales: shoulder/arm (0-36), wrist/hand (0-24), coordination (0-6). Higher scores indicate better function. Units on a scale.
Time Frame: Retention of measure comparing baseline to one-month post training
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | START
Number analyzed (Participants) | 11 | 10
units on a scale | -0.5 (5.291503) | -0.333333 (5.715476)

7. Secondary Outcome: Change in Stroke Impact Scale From Baseline to Post-intervention
Description: The Stroke Impact Scale (SIS) measures quality of life and functional recovery post-stroke across 8 subscales: strength (0-100), hand function (0-100), mobility (0-100), ADL (0-100), emotion (0-100), memory (0-100), communication (0-100), participation (0-100). Each subscale score is scaled to 0-100; higher scores indicate better outcomes. The total score (0-100) averages the subscale scores. Change in total score is reported. Units on a scale.
Time Frame: Change from baseline to post-intervention (1 week intervention, 1 month post intervention - total 5 weeks time frame)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | START
Number analyzed (Participants) | 11 | 10
units on a scale | 0.363636 (2.01359) | -0.777778 (1.922094)

8. Secondary Outcome: Retention of Stroke Impact Scale - Post-training to One-month Post
Description: as for outcome 7
Time Frame: Change from baseline to one-month post training
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | START
Number analyzed (Participants) | 11 | 10
units on a scale | -1.375 (1.685018) | 2.5 (3.391165)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at the conclusion of the experiment, with no long-term monitoring conducted. The total duration was 5 weeks of monitoring from start (Baseline) to end of experiment (one month post intervention)
Description: There were no adverse events.
Groups:
- Control: The control group received standard care without additional intervention. Participants underwent routine medical management and assessments as per the trial protocol, serving as a comparator to evaluate the START intervention's effects.
- Start - Intervention: The START intervention group received the Stroke Therapy and Rehabilitation Training (START) program, a targeted upper extremity rehabilitation protocol. This included structured exercises to improve motor function, delivered alongside standard care, with outcomes compared to the control group.
Arm/Group | Control | Start - Intervention
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

LIMITATIONS AND CAVEATS:
This trial was ended early as preliminary data assessed that it would not be successful. PI indicates that clinical assessment measures may not have been sensitive to pick up the small changes that the PI has previously picked up. Further, the trial was only 3 days in length and longer may be required to see changes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT05277389/Prot_SAP_ICF_000.pdf